CLINICAL TRIAL: NCT02858232
Title: A Single Arm, Open, Phase I/II Clinical Study of MASCT-I Treatment for Advanced Solid Tumor
Brief Title: MASCT-I Treatment for Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: Hengrui Yuanzheng Bio-Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LYG1602-01-02
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Solid Tumors
Keywords: MASCT-I; Solid Tumors

ARMS (1):
- solid tumor (Experimental): Multiple Target Antigen Stimulating Cell Therapy (MASCT-I)
  Interventions: Biological: MASCT-I

INTERVENTIONS:
Biological: MASCT-I — Dendritic cells(DC) loaded with antigens ih day 8, cytotoxic T lymphocytes ( CTL) induced by DC IV day 21-28, every 28 days until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Other Names: Multiple Target Antigen Stimulating Cell Therapy

SUMMARY:
Multiple Target Antigen Stimulating Cell Therapy (MASCT-I) is a new immunotherapy that dendritic cells(DC) was induced from autologous peripheral blood. The DC can then be loaded with antigens and re-infused. In vitro, antigen-pulsed DC can stimulate autologous T-cell proliferation and induction of autologous specific cytotoxic T-cells(CTL)，similarly re-infused. The previous research data showed that MASCT had the modest overall response and less adverse effects for Hepatocellular Carcinoma patients.

The study is aimed to evaluate the safety of MASCT-1 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is divided into two stages. The first stage is the safety study in small samples, and the second stage is the sample size expansion phase.

40-50 patients with advanced or recurrent solid tumors who had failed after standard treatment will be recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed, advanced (unresectable) solid tumors（Lung cancer, colon cancer, prostate cancer, soft tissue sarcoma, other rare tumor） who have progressed on standard therapy.
2. With written informed consent signed voluntarily by patients themselves.
3. The time of between Patients enrollment and the end of other anti-tumors therapies≥1 month.
4. ECOG≤2.
5. At least one measurable lesion as defined by RECIST criteria 1.1 for tumors.
6. Life expectancy ≥6 months.
7. With normal cardiopulmonary function.
8. Patients have adequate organ function as defined by the following criteria:

Hemoglobin (HGB) ≥85g/L Absolute neutrophil count (ANC) ≥1.0×10^9/L White blood cell (WBC) ≥3.0×10^9/L Platelet count ≥80×10^9/L Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) of ≤2.5 upper normal limitation (UNL) or ≤5 UNL in case of liver metastasis Alkaline phosphatase (ALP)≤2.5 UNL Total bilirubin (TBil) of ≤1.5 UNL Blood urea nitrogen (BUN) and Creatinine (Cr) of≤1.5 UNL Albumin (ALB) ≥30g/L

Exclusion Criteria:

1. Pregnant or expecting to pregnant
2. Participated in other clinical trials before screening except of observational study.
3. Refused to provide blood samples.
4. Known allergic history of sodium citrate drugs.
5. Known history of organ transplant, including autologous bone marrow transplantation and peripheral stem cell transplantation.
6. Known active brain metastases
7. The use of immunosuppressive drugs with current or 14 days before enrollment.
8. Active primary immune deficiency.
9. known history of tuberculosis.
10. Active infection, including hepatitis B, hepatitis C virus, or human immunodeficiency virus.
11. Patients with serious infection, hepatopathy, nephropathy, respiratory disease, cardiovascular disease or incontrollable diabetes, etc.
12. Patients have other malignant tumors within 5 years,excluding melanoma and carcinoma in situ of cervix.
13. Clinical signs of heart disease.
14. Treatment with any anti-tumors agent within 28days of first administration of study treatment.
15. The research on the influence of non legal persons, medical or ethical reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | up to 2 years
  The incidence of treatment-related adverse events were graded with the use of the National Cancer Institute Common Terminology Criteria for Adverse Events, versio4.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  clinical response of treatment according to RESIST v1.1 criteria
Disease Control Rate (DCR) | up to 2 years
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) based on RESIST v1.1 criteria.
Progression-Free Survival (PFS) | From enrollment to progression of disease. Estimated about 6 months
  The length of time from enrollment until the time of progression of disease
Overall Survival (OS) | up to 2 years
  From enrollment to death of patients

OTHER OUTCOMES:
The relationship between clinical efficacy and antigen specific immune response | up to 2 years